CLINICAL TRIAL: NCT04889040
Title: A Multicenter, Phase III Randomized, Double-Blind, Placebo-Controlled, Outpatient Study to Evaluate the Efficacy, Safety, Antiviral Activity of RO7496998 (AT-527) in Patients With Mild or Moderate COVID-19
Brief Title: Study to Evaluate the Effects of RO7496998 (AT-527) in Non-Hospitalized Adult and Adolescent Participants With Mild or Moderate COVID-19
Acronym: MORNINGSKY
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on program revaluation and in agreement with the co-development partner the sponsor took the decision to terminate this study.
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV43043; 2020-005759-18 (EudraCT Number); NCT05126576 (obsolete NCT alias)
Record Dates: First submitted 2021-05-10; First posted 2021-05-17 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
Keywords: Coronavirus Disease 2019; COVID-19; antiviral drug; SARS-CoV-2; Mild to Moderate COVID-19; antiviral efficacy
MeSH Terms: conditions — COVID-19 | interventions — AT-511

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): The dose and regimen of the placebo will match that of AT-527.
  Interventions: Drug: Placebo
- RO7496998 (AT-527) (Experimental): Orally administered, 550 mg twice daily (BID) for 5 days
  Interventions: Drug: RO7496998

INTERVENTIONS:
Drug: RO7496998 — 275 mg tablets
  Other Names: AT-527
  Arms: RO7496998 (AT-527)
Drug: Placebo — Matching tablets
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy, safety, antiviral activity, and pharmacokinetics of study drug RO7496998 (AT-527) compared to placebo in non-hospitalized adult and adolescent participants with mild to moderate coronavirus disease 2019 (COVID-19) in the outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Positive SARS-CoV-2 diagnostic test (RT-PCR or validated rapid antigen test) ≤72 hours prior to randomization
* At least three of the following symptoms of at least moderate (score ≥2 as per COVID-19 Symptom Diary) intensity: nasal congestion or runny nose, sore throat, cough, shortness of breath, muscle or body aches, fatigue, headache, chills or sweats, feeling hot or feverish, nausea, vomiting, or diarrhea.
* Has symptoms consistent with mild or moderate COVID-19, as determined by the investigator, with onset ≤5 days before dosing on Day 1

Exclusion Criteria:

* Clinical signs indicative of COVID-19 illness requiring hospitalization
* Admitted to a hospital prior to randomization or is hospitalized (inpatient) at randomization due to COVID-19
* In the opinion of the investigator, is likely to experience imminent deterioration and require hospitalization
* Treatment with an investigational drug within 5 half-lives or 3 months (whichever is longer) of randomization
* Treatment with a COVID-19 therapeutic agent including, but not limited to, other direct or indirect acting antivirals against SARS-CoV-2 (such as remdesivir or favipiravir), systemic or inhaled steroids (such as dexamethasone or inhaled budesonide), colchicine, ivermectin, interferons, convalescent plasma, monoclonal antibodies against SARS CoV-2 or interleukin 6 (IL-6), intravenous immunoglobulin or other EUA-approved treatments within 3 months or less than 5 drug elimination half-lives (whichever is longer) prior to the screening visit
* Concomitant use of P-glycoprotein inhibitors or inducers listed as prohibited therapy in the protocol
* Known allergy or hypersensitivity to components of study drug
* Abnormal laboratory test results at screening
* Requirement of any prohibited medications during the study
* Other known active viral or bacterial infection at the time of screening, such as influenza
* Any clinically significant medical condition or laboratory abnormality that, in the opinion of the investigator, could jeopardize the safety of the patient or affect patient compliance or safety/efficacy observations during the study
* COVID-19 vaccination within ≤ 40-days prior to enrollment (second dose if applicable)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (50):
- Instituto Ave Pulmo, Mar del Plata, Argentina
- Belgium (3):
  - Maison Médicale La Brèche, Châtelineau
  - Private Practice Dr Jean Benoit Martinot, Erpent
  - Medif, Gozée
- Brazil (5):
  - L2 Ip Instituto de Pesquisas Clinicas Ltda ME; Centro Medico Hospitalar, Brasília, Federal District
  - Chronos Pesquisa Clinica, Taguatinga, Federal District
  - Hospital Nossa Senhora das Graças, Curitiba, Paraná
  - Hospital Agamenon Magalhães, Recife, Pernambuco
  - Conjunto Hospitalar do Mandaqui, São Paulo, São Paulo
- Denmark (2):
  - Aalborg Universitetshospital, Aalborg
  - Rigshospitalet Copenhagen University Hospital, Copenhagen
- Praxis am Ebertplatz, Cologne, Germany
- Japan (13):
  - Higashiosaka city Medical Center, Higashiosaka-Shi
  - Rinku General Medical Center, Izumisano
  - Sagamihara Kyodo Hospital, Kanagawa
  - Misyuku hospital, Meguro-Ku
  - IUHW Narita Hospital, Narita
  - Houjin Syadan Kouhoukai Takagi Hospital, Okawa-Shi
  - Okayama City Hospital, Okayama
  - Ome Municipal General Hospital, Ome-Shi
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakaishi
  - Tokyo Shinagawa Hospital Medical Corporation Association Tokyokyojuno-kai, Shinagawa City
  - Edogawa Medicare Hospital, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine, Tokyo
  - Tokyo Medical University Hachioji Medical Center, Tokyo
- Mexico (6):
  - CIMAB SA de CV, Torreón, Coahuila
  - Panamerican Clinical Research S.A de C.V., Guadalajara, Jalisco
  - Clinstile S.A de C.V., Mexico City, Mexico CITY (federal District)
  - PanAmerican Clinical Research, Querétaro, Queréaro, Querétaro
  - Instituto Jalisciense de Investigacion Clinica S.A. de C.V., Guadalajara
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, México
- Unidade Local de Saude de Matosinhos SA, Matosinhos Municipality, Portugal
- Romania (3):
  - Prof. Dr. Matei Bals Institute of Infectious Diseases, Bucharest
  - County Hospital Caracal, Caracal
  - Sibiu Emergency Clinical County Hospital, Sibiu
- Switzerland (2):
  - Hôpital Universitaire de Genève (HUG), Geneva
  - Universitätsspital Zürich, Zurich
- Turkey (Türkiye) (4):
  - Gazi Universitesi Tip Fakultesi, Ankara
  - Ankara University Medical Faculty - PPDS, Çankaya
  - Ege University Medical Faculty, Izmir
  - Karadeniz Technical University Faculty of Medicine, Trabzon
- Ukraine (9):
  - Municipal Non-profit Enterprise ?City Clinical Hospital #13? of Kharkiv City Council, Kharkiv, Kharkiv Governorate
  - Public Non-Profit Enterprise ?City Outpatient Clinic #9? of Kharkiv City Council, Kharkiv, Kharkiv Governorate
  - CNPE City Clinical Hospital #6 of DCC, Dnipro, Kholm Governorate
  - Medical Center LLC "Harmony of Beauty", Kyiv, KIEV Governorate
  - CNE Kyiv City Clinical Hospital#1 of Exec. Body, Kyiv, KIEV Governorate
  - Kyiv Railway Clinical Hospital No2 of Branch Health Center of the JSC Ukrainian Rail, Kyiv, KIEV Governorate
  - Polyclinic of Center of Medical Service and Rehabilitation of State JSHC Artem, Kyiv, KIEV Governorate
  - Communal Non-Commercial Enterprise Vinnytsia City Clinical Hospital 1, Vinnytsia, Podolia Governorate
  - Communal Non-Profit Enterprise City Hospital #7 of Zaporizhzhia City Council, Zaporizhzhia, Tavria Okruha

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm)

REFERENCES:
- [Derived] Horga A, Saenz R, Yilmaz G, Simon-Campos A, Pietropaolo K, Stubbings WJ, Collinson N, Ishak L, Zrinscak B, Belanger B, Granier C, Lin K, C Hurt A, Zhou XJ, Wildum S, Hammond J. Oral bemnifosbuvir (AT-527) vs placebo in patients with mild-to-moderate COVID-19 in an outpatient setting (MORNINGSKY). Future Virol. 2023 Oct:10.2217/fvl-2023-0115. doi: 10.2217/fvl-2023-0115. Epub 2023 Nov 1. PMID 37928891

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were non-hospitalized, with mild to moderate COVID-19, with or without risk factors for severe disease.
Period: Overall Study
Arm/Group | Placebo | RO7496998 (AT-527)
Started | 73 | 143
Received Treatment | 71 | 141
Completed | 68 | 138
Not Completed | 5 | 5
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | RO7496998 (AT-527) | Total
Number analyzed (Participants) | 73 | 143 | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (14.9) | 41.1 (13.2) | 41.3 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 62 | 94
  Male | 41 | 81 | 122
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 9 | 15
  Asian | 14 | 26 | 40
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 3 | 4
  White | 50 | 105 | 155
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Number of COVID-19 Symptoms Present at Baseline [Mean (Standard Deviation); unit: Number of Covid-19 Symptoms] — Population: All participants who were randomized to treatment, received a dose of study treatment, were reverse transcriptase quantitative polymerase chain reaction (RT-qPCR) positive for SARS-CoV-2 at any point during the study and did not have missing data.
  Number of Covid-19 Symptoms
    number analyzed (Participants) | 68 | 130 | 198
    (all) | 7.85 (2.58) | 7.92 (2.74) | 7.90 (2.68)

OUTCOME MEASURES:

1. Primary Outcome: Time to Alleviation or Improvement of COVID-19 Symptoms (21.5 Hours)
Description: COVID-19 symptoms will be evaluated using the COVID-19 Symptom Diary (questions 1-12). The severity of each COVID-19 symptom will be recorded on a Likert scale (i.e none/mild/moderate/severe).
  The time to alleviation or improvement of COVID-19 symptoms is defined as follows: for new symptoms, it is defined as the length of time taken from randomization to the point at which a Score of 0 or 1 has been maintained for a duration of at least 21.5 hours. For preexisting symptoms, it is defined as the time from randomization to when a patient's symptoms have been maintained or improved (requires at least a single category improvement from baseline on the COVID-19 Symptom Diary Likert scale) for a duration of 21.5 hours.
Time Frame: Up to 29 days
Population: All participants who were randomized to treatment, received a dose of study treatment, and were RT-qPCR positive for SARS-CoV-2 at any point during the study.
Measure: Median (97.5% Confidence Interval); unit: hours
Arm/Group | Placebo | RO7496998 (AT-527)
Number analyzed (Participants) | 70 | 137
hours | 73.7 [47.1 to 105.8] | 94.5 [68.1 to 131.7]

2. Secondary Outcome: Time to Alleviation or Improvement of COVID-19 Symptoms (43 Hours)
Description: COVID-19 symptoms will be evaluated using the COVID-19 Symptom Diary (questions 1-12). The severity of each COVID-19 symptom will be recorded on a Likert scale (i.e none/mild/moderate/severe).
  The time to alleviation or improvement of COVID-19 symptoms is defined as follows: for new symptoms, it is defined as the length of time taken from randomization to the point at which a Score of 0 or 1 has been maintained for a duration of at least 43 hours. For preexisting symptoms, it is defined as the time from randomization to when a patient's symptoms have been maintained or improved (requires at least a single category improvement from baseline on the COVID-19 Symptom Diary Likert scale) for a duration of 43 hours.
Time Frame: Up to 29 days
Population: as for outcome 1
Measure: Median (97.5% Confidence Interval); unit: hours
Arm/Group | Placebo | RO7496998 (AT-527)
Number analyzed (Participants) | 70 | 137
hours | 79.6 [55.7 to 108.2] | 109.5 [83.8 to 147.5]

3. Secondary Outcome: Time to Alleviation of COVID-19 Symptoms (21.5 Hours)
Description: Time from randomization to the point at which the following criterion is met and maintained for at least 21.5 hours.
  - Score of 0 or 1 on Items 1-12 of the COVID-19 Symptom Diary.
Time Frame: Up to 29 days
Population: as for outcome 1
Measure: Median (97.5% Confidence Interval); unit: hours
Arm/Group | Placebo | RO7496998 (AT-527)
Number analyzed (Participants) | 70 | 137
hours | 73.7 [47.1 to 105.8] | 94.5 [68.1 to 131.7]

4. Secondary Outcome: Time to Alleviation of COVID-19 Symptoms (43 Hours)
Description: Time from randomization to the point at which the following criterion is met and maintained for at least 43 hours.
  - Score of 0 or 1 on Items 1-12 of the COVID-19 Symptom Diary.
Time Frame: Up to 29 days
Population: as for outcome 1
Measure: Median (97.5% Confidence Interval); unit: hours
Arm/Group | Placebo | RO7496998 (AT-527)
Number analyzed (Participants) | 70 | 137
hours | 79.6 [55.7 to 108.2] | 109.5 [83.8 to 147.5]

5. Secondary Outcome: Time to One-Category Improvement of Baseline Presenting COVID-19 Symptoms
Description: Time from randomization to the point at which symptoms (Items 1-12 of the COVID-19 Symptom Diary) have improved by at least one category from baseline on the COVID-19 Symptom Diary Likert scale, maintained for at least 21.5 hours.
Time Frame: Up to 29 days
Population: All participants who were randomized to treatment, received a dose of study treatment, were RT-qPCR positive for SARS-CoV-2 at any point during the study and with baseline symptoms.
Measure: Median (97.5% Confidence Interval); unit: hours
Arm/Group | Placebo | RO7496998 (AT-527)
Number analyzed (Participants) | 68 | 130
hours | 70.9 [41.8 to 91.8] | 81.5 [60.5 to 119.9]

6. Secondary Outcome: Time to Alleviation of Individual Symptoms
Description: Time from randomization to the point at which the following criterion is met and maintained (for each individual symptom) for at least 21.5 hours.
  - Score of 0 or 1 for Items 1-14 of the COVID-19 Symptom Diary
Time Frame: Up to 29 days
Population: All participants who were randomized to treatment, received a dose of study treatment, were RT-qPCR positive for SARS-CoV-2 at any point during the study and had a symptom score of >= 2 at baseline.
Measure: Median (97.5% Confidence Interval); unit: hours
Arm/Group | Placebo | RO7496998 (AT-527)
Number analyzed (Participants) | 70 | 137
hours
  Nasal Congestion or Runny Nose: number analyzed (Participants) | 36 | 65
  Nasal Congestion or Runny Nose | 36.4 [23.4 to 60.6] | 37.3 [23.4 to 57.6]
  Sore Throat: number analyzed (Participants) | 19 | 43
  Sore Throat | 45.6 [23.4 to 75.1] | 33.2 [20.9 to 54.3]
  Cough: number analyzed (Participants) | 33 | 55
  Cough | 37.6 [26.8 to 118.7] | 49.5 [28.4 to 106.4]
  Shortness of Breath: number analyzed (Participants) | 12 | 14
  Shortness of Breath | 24.0 [11.8 to 106.8] | 47.5 [32.4 to 96.8]
  Muscle or Body Aches: number analyzed (Participants) | 27 | 59
  Muscle or Body Aches | 35.3 [14.3 to 59.4] | 44.9 [33.1 to 53.0]
  Fatigue: number analyzed (Participants) | 32 | 70
  Fatigue | 66.6 [36.5 to 118.9] | 61.3 [47.1 to 108.1]
  Headache: number analyzed (Participants) | 20 | 53
  Headache | 23.2 [14.5 to 41.8] | 41.4 [24.4 to 59.5]
  Chills/Sweats: number analyzed (Participants) | 25 | 52
  Chills/Sweats | 36.0 [22.5 to 57.6] | 39.0 [28.4 to 50.5]
  Feeling Hot or Feverish: number analyzed (Participants) | 18 | 40
  Feeling Hot or Feverish | 24.6 [16.4 to 66.7] | 36.2 [19.7 to 61.4]
  Nausea: number analyzed (Participants) | 2 | 11
  Nausea | 31.4 [11.1 to NA] — Not evaluable due to an insufficient number of events | 43.5 [22.6 to 73.4]
  Vomiting: number analyzed (Participants) | 2 | 1
  Vomiting | 20.1 [16.4 to NA] — Not evaluable due to an insufficient number of events | 33.0 [NA to NA] — Not evaluable due to an insufficient number of events
  Diarrhea: number analyzed (Participants) | 9 | 10
  Diarrhea | 17.6 [14.9 to 73.6] | 66.7 [19.8 to 107.2]
  Sense of Smell: number analyzed (Participants) | 21 | 37
  Sense of Smell | 132.6 [84.3 to 229.0] | 104.9 [72.6 to 206.0]
  Sense of Taste: number analyzed (Participants) | 17 | 21
  Sense of Taste | 128.9 [84.3 to 202.2] | 155.7 [52.5 to 371.7]

7. Secondary Outcome: Percentage of Participants Requiring Hospitalization for COVID-19
Description: Hospitalizations for COVID-19 are defined as SAEs for which the investigator has cited that the suspected cause was the disease under study and where there is a non-missing hospital admission date.
Time Frame: Up to Day 33 visit
Population: as for outcome 1
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | RO7496998 (AT-527)
Number analyzed (Participants) | 70 | 137
percentage of participants | 10.0 [1.25 to 18.75] | 2.9 [0.00 to 6.51]

8. Secondary Outcome: Percentage of Participants With Greater Than or Equal to 1 COVID-19 Related Medically Attended Visit
Description: Medically attended visit is defined as hospitalization, emergency room (ER) visit, urgent care visit, physician's office visit, or telemedicine visit, with the primary reason for the visit being COVID-19.
Time Frame: Up to Day 33 visit
Population: as for outcome 1
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | RO7496998 (AT-527)
Number analyzed (Participants) | 70 | 137
percentage of participants | 14.3 [4.20 to 24.37] | 10.2 [4.05 to 16.38]

9. Secondary Outcome: Duration of Fever
Description: Time to return to an afebrile state (temperature ≤ 37.5°C) maintained for at least 21.5 hours.
Time Frame: Up to 29 days
Population: All participants who were randomized to treatment, received a dose of study treatment, were RT-qPCR positive for SARS-CoV-2 at any point during the study, and had a fever at baseline.
Measure: Median (97.5% Confidence Interval); unit: hours
Arm/Group | Placebo | RO7496998 (AT-527)
Number analyzed (Participants) | 12 | 20
hours | 47.3 [12.6 to 82.2] | 55.7 [25.9 to 96.4]

10. Secondary Outcome: Percentage of Participants With COVID-19 Related Complications
Description: COVID-related complications are defined as death, hospitalization, pneumonia, sepsis, coagulopathy, pericarditis/myocarditis and cardiac failure.
  Pneumonia, acute respiratory failure, sepsis, coagulopathy, pericarditis/myocarditis, and cardiac failure were adjudicated per blinded manual medical review of events by an internal adjudication team before study readout.
Time Frame: Up to Day 33 visit
Population: as for outcome 1
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | RO7496998 (AT-527)
Number analyzed (Participants) | 70 | 137
percentage of participants | 10.0 [1.25 to 18.75] | 4.4 [0.10 to 8.66]

11. Secondary Outcome: Percentage of Participants With Any Post-Treatment Infection
Description: Post-treatment infections were defined as any treatment-emergent adverse event with a primary system organ class of infections and infestations.
Time Frame: Up to Day 33 visit
Population: as for outcome 1
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | RO7496998 (AT-527)
Number analyzed (Participants) | 70 | 137
percentage of participants | 14.3 [4.20 to 24.37] | 9.5 [3.51 to 15.47]

12. Secondary Outcome: Change From Baseline in the Amount of Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) Virus RNA
Description: SARS-CoV-2 virus RNA will be measured by reverse-transcriptase quantitative polymerase chain reaction (RT-qPCR)
Time Frame: Baseline and on Days 3, 5, 7 and 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Placebo | RO7496998 (AT-527)
Number analyzed (Participants) | 70 | 137
log10 copies/mL
  Baseline: number analyzed (Participants) | 69 | 137
  Baseline | 6.49 (1.61) | 6.59 (1.54)
  Day 3: number analyzed (Participants) | 68 | 137
  Day 3 | -1.05 (1.06) | -1.07 (1.16)
  Day 5: number analyzed (Participants) | 67 | 136
  Day 5 | -2.24 (1.40) | -2.01 (1.50)
  Day 7: number analyzed (Participants) | 66 | 135
  Day 7 | -3.10 (1.38) | -2.98 (1.66)
  Day 14: number analyzed (Participants) | 65 | 128
  Day 14 | -4.21 (1.64) | -4.25 (1.64)

13. Secondary Outcome: Time to Cessation of SARS-CoV-2 Viral Shedding
Description: Defined as time from randomization to the first time when a negative qualitative virus RNA by RT-PCR test result is obtained.
Time Frame: Up to 14 days
Population: as for outcome 1
Measure: Median (97.5% Confidence Interval); unit: days
Arm/Group | Placebo | RO7496998 (AT-527)
Number analyzed (Participants) | 70 | 137
days | 13.0 [12.8 to NA] — Not evaluable due to an insufficient number of events | 13.0 [13.0 to 13.1]

14. Secondary Outcome: Percentage of Participants Positive for SARS-CoV-2 Virus RNA at Specified Timepoints
Description: Defined as percentage of participants with a positive qualitative virus RNA by RT-PCR.
Time Frame: Baseline and on Days 3, 5, 7 and 14
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | RO7496998 (AT-527)
Number analyzed (Participants) | 70 | 137
percentage of participants
  Baseline: number analyzed (Participants) | 69 | 137
  Baseline | 97.1 | 100
  Day 3: number analyzed (Participants) | 68 | 137
  Day 3 | 98.5 | 96.4
  Day 5: number analyzed (Participants) | 68 | 136
  Day 5 | 89.7 | 91.9
  Day 7: number analyzed (Participants) | 67 | 135
  Day 7 | 74.6 | 76.3
  Day 14: number analyzed (Participants) | 66 | 128
  Day 14 | 43.9 | 34.4

15. Secondary Outcome: Area Under the Curve (AUC) in the Amount of SARS-CoV-2 Virus RNA
Time Frame: Day 1 prior to dosing, Day 3, Day 5, Day 7 and Day 14
Population: All participants who were randomized to treatment, received a dose of study treatment, were RT-qPCR positive for SARS-CoV-2 at any point during the study, and had at least 2 or more virology assessments.
Measure: Mean (Standard Deviation); unit: log10 copies/mL*hour
Arm/Group | Placebo | RO7496998 (AT-527)
Number analyzed (Participants) | 69 | 137
log10 copies/mL*hour | 1122.39 (339.70) | 1174.30 (377.49)

16. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Time Frame: Up to Day 33 visit
Population: All participants who received at least one dose of study treatment
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | RO7496998 (AT-527)
Number analyzed (Participants) | 71 | 141
percentage of participants | 36.6 | 39.0

17. Secondary Outcome: Plasma Concentration of AT-511 at Specified Timepoints
Description: AT-511 is the free base form of RO7496998 (AT-527).
Time Frame: Up to 7 days
Population: All participants who received AT-527 and had at least one post-dose drug concentration measurement at a scheduled visit time point
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | RO7496998 (AT-527)
Number analyzed (Participants) | 137
nanograms per milliliter (ng/mL)
  Day 1, 0 hour: number analyzed (Participants) | 133
  Day 1, 0 hour | 17.4 (158.6)
  Day 1, 1 hour: number analyzed (Participants) | 136
  Day 1, 1 hour | 1456.8 (1757.7)
  Day 1, 2 hours: number analyzed (Participants) | 5
  Day 1, 2 hours | 1029.3 (1085.5)
  Day 1, 4 hours: number analyzed (Participants) | 5
  Day 1, 4 hours | 206.3 (289.5)
  Day 5, 0 hour: number analyzed (Participants) | 125
  Day 5, 0 hour | 52.8 (271.0)
  Day 5, 1 hour: number analyzed (Participants) | 125
  Day 5, 1 hour | 1659.0 (2213.9)
  Day 5, 2 hours: number analyzed (Participants) | 4
  Day 5, 2 hours | 1934.5 (2210.6)
  Day 5, 4 hours: number analyzed (Participants) | 4
  Day 5, 4 hours | 202.3 (310.7)
  Day 5, 8 hours: number analyzed (Participants) | 4
  Day 5, 8 hours | 8.8 (9.5)
  Day 5, 48 hours: number analyzed (Participants) | 129
  Day 5, 48 hours | 4.6 (40.9)

18. Secondary Outcome: Plasma Concentration of AT-551 at Specified Timepoints
Description: AT-511 is the free base form of RO7496998 (AT-527). Major metabolites are AT-551, AT-229, and AT-273 (a surrogate for the intracellular concentration of the active triphosphate metabolite AT-9010)
Time Frame: Up to 7 days
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | RO7496998 (AT-527)
Number analyzed (Participants) | 137
nanograms per milliliter (ng/mL)
  Day 1, 0 hour: number analyzed (Participants) | 133
  Day 1, 0 hour | 1.9 (12.2)
  Day 1, 1 hour: number analyzed (Participants) | 135
  Day 1, 1 hour | 166.9 (209.8)
  Day 1, 2 hours: number analyzed (Participants) | 5
  Day 1, 2 hours | 335.7 (257.6)
  Day 1, 4 hours: number analyzed (Participants) | 5
  Day 1, 4 hours | 195.0 (146.4)
  Day 5, 0 hour: number analyzed (Participants) | 125
  Day 5, 0 hour | 49.1 (65.0)
  Day 5, 1 hour: number analyzed (Participants) | 125
  Day 5, 1 hour | 150.2 (144.5)
  Day 5, 2 hours: number analyzed (Participants) | 4
  Day 5, 2 hours | 213.6 (201.7)
  Day 5, 4 hours: number analyzed (Participants) | 4
  Day 5, 4 hours | 138.8 (136.2)
  Day 5, 8 hours: number analyzed (Participants) | 4
  Day 5, 8 hours | 27.5 (17.5)
  Day 5, 48 hours: number analyzed (Participants) | 129
  Day 5, 48 hours | 2.6 (5.2)

19. Secondary Outcome: Plasma Concentration of AT-229 at Specified Timepoints
Description: as for outcome 18
Time Frame: Up to 7 days
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | RO7496998 (AT-527)
Number analyzed (Participants) | 137
nanograms per milliliter (ng/mL)
  Day 1, 0 hour: number analyzed (Participants) | 133
  Day 1, 0 hour | 2.2 (18.4)
  Day 1, 1 hour: number analyzed (Participants) | 135
  Day 1, 1 hour | 123.6 (172.5)
  Day 1, 2 hours: number analyzed (Participants) | 5
  Day 1, 2 hours | 507.8 (497.5)
  Day 1, 4 hours: number analyzed (Participants) | 5
  Day 1, 4 hours | 354.4 (259.2)
  Day 5, 0 hour: number analyzed (Participants) | 125
  Day 5, 0 hour | 367.8 (259.1)
  Day 5, 1 hour: number analyzed (Participants) | 125
  Day 5, 1 hour | 418.0 (257.6)
  Day 5, 2 hours: number analyzed (Participants) | 4
  Day 5, 2 hours | 454.3 (331.7)
  Day 5, 4 hours: number analyzed (Participants) | 4
  Day 5, 4 hours | 490.1 (296.4)
  Day 5, 8 hours: number analyzed (Participants) | 4
  Day 5, 8 hours | 279.6 (176.0)
  Day 5, 48 hours: number analyzed (Participants) | 129
  Day 5, 48 hours | 118.7 (127.2)

20. Secondary Outcome: Plasma Concentration of AT-273 at Specified Timepoints
Description: as for outcome 18
Time Frame: Up to 7 days
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | RO7496998 (AT-527)
Number analyzed (Participants) | 137
nanograms per milliliter (ng/mL)
  Day 1, 0 hour: number analyzed (Participants) | 133
  Day 1, 0 hour | 0.7 (2.5)
  Day 1, 1 hour: number analyzed (Participants) | 135
  Day 1, 1 hour | 15.5 (26.9)
  Day 1, 2 hours: number analyzed (Participants) | 5
  Day 1, 2 hours | 135.1 (136.2)
  Day 1, 4 hours: number analyzed (Participants) | 5
  Day 1, 4 hours | 173.5 (120.6)
  Day 5, 0 hour: number analyzed (Participants) | 125
  Day 5, 0 hour | 149.8 (78.1)
  Day 5, 1 hour: number analyzed (Participants) | 125
  Day 5, 1 hour | 141.7 (72.7)
  Day 5, 2 hours: number analyzed (Participants) | 4
  Day 5, 2 hours | 108.8 (61.0)
  Day 5, 4 hours: number analyzed (Participants) | 4
  Day 5, 4 hours | 172.7 (129.2)
  Day 5, 8 hours: number analyzed (Participants) | 4
  Day 5, 8 hours | 118.6 (80.2)
  Day 5, 48 hours: number analyzed (Participants) | 129
  Day 5, 48 hours | 48.4 (32.7)

ADVERSE EVENTS:
Time Frame: up to the Day 33 visit
Description: Safety analyses were performed on the safety evaluable set, which consisted of all randomized participants who received at least one dose of study treatment.
Groups:
- AT-527: Orally administered, 550 mg twice daily (BID) for 5 days
Arm/Group | Placebo | AT-527
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/141
Serious Adverse Events (participants affected / at risk) | 7/71 | 5/141
Other Adverse Events (participants affected / at risk) | 5/71 | 11/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=71) | AT-527 (N=141)
COVID-19 (Infections and infestations) | 3 (3) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 4 (4) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=71) | AT-527 (N=141)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 8 (8)
Headache (Nervous system disorders) | 5 (5) | 4 (4)

LIMITATIONS AND CAVEATS:
The study was terminated with only 16% of the planned sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT04889040/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/40/NCT04889040/SAP_001.pdf